CLINICAL TRIAL: NCT01788436
Title: An Exploratory Study to Measure and Contrast Implicit and Explicit Learning Performance in Patients With Stable Schizophrenia and Young and Elderly Healthy Subjects
Brief Title: A Study to Assess Learning Performance in Patients With Schizophrenia and Young and Elderly Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CR100911; NOCOMPOUNDEDI0004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-11-08; First posted 2013-02-11 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Young healthy volunteers; Elderly healthy volunteers; Learning performance
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Patients with schizophrenia (Experimental)
  Interventions: Behavioral: Cognitive Test Battery 1; Behavioral: Cognitive Test Battery 2
- Group 2: Young healthy volunteers (Active Comparator)
  Interventions: Behavioral: Cognitive Test Battery 1; Behavioral: Cognitive Test Battery 2
- Group 3: Elderly healthy volunteers (Experimental)
  Interventions: Behavioral: Cognitive Test Battery 1; Behavioral: Cognitive Test Battery 2

INTERVENTIONS:
Behavioral: Cognitive Test Battery 1 — The Cognitive Test Battery 1 comprises the following tasks: Practice with graphics tablet, pen and screen; Digit Symbol Substitution Test (DSST); Implicit Pattern/Sequence Learning Task (PLT_Impl); Verbal Learning Test (VLT); Figure drawing; Mirror Drawing; Explicit Pattern Learning Task (PLT_Expl); Delayed Recall and Recognition Test; and Pursuit rotor.
Behavioral: Cognitive Test Battery 2 — The Cognitive Test Battery 2 comprises the following tasks: Practice with graphics tablet, pen and screen; Digit Symbol Substitution Test (DSST); Implicit Learning Retention Test; Hopkins Verbal Learning Test (HVLT); Figure drawing; Mirror Drawing; Explicit Learning Retention Test; Instrumental Learning Task; Pursuit rotor; and Sensory Motor Interception Adaptation Task.

SUMMARY:
The purpose of this study is to measure and contrast implicit and explicit learning performance in patients with schizophrenia relative to young and elderly healthy volunteers.

DETAILED DESCRIPTION:
This is an exploratory study involving schizophrenic patients (Group 1) and young and elderly healthy volunteers (Group 2 and 3 respectively). No investigational medicinal product will be administered. For all participants enrolled (Group 1 to 3) the study will consist of an eligibility screening examination (from Day -21 up to and including Day 1) and 3 cognitive assessment days. Cognitive assessments will be made on 2 subsequent days (Days 1 and 2) which are separated by overnight sleep. In addition, a session will be performed on Day 7. Completion of the cognitive test batteries can occur at any time during the day provided that the completion time is comparable on all test days. For each participant, the maximal study duration will not exceed 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (patients with schizophrenia):
* Be a man or woman between 18 and 55 years of age, inclusive
* Has a known history of schizophrenia of at least 12 months by the referring psychiatrist
* Receives stable antipsychotic drug therapy (maximally 2) for at least 6 weeks prior to screening
* Medically stable on the basis of clinical judgment by the investigator
* Group 2 (young healthy volunteers): be a healthy man or woman between 18 and 55 years of age, inclusive
* Group 3 (elderly healthy volunteers): be a healthy man or woman between 65 and 85 years of age, inclusive
* All participants (Group 1 to 3) must be capable of completing the cognitive test battery

Exclusion Criteria:

* Receives treatment with benzodiazepines, tricyclic antidepressant or anticholinergics
* Has a positive urine screen for drugs of abuse or alcohol breath test
* Has a recent history (within previous 6 months) of alcohol or drug abuse
* Has psychological and/or emotional problems, which would render the informed consent invalid, or limit the ability of the participant to comply with the study requirements
* Has any condition that, in the opinion of the investigator, would compromise the wellbeing of the participant or the study or prevent the participant from meeting or performing study requirements
* Group 1 only: a diagnosis of substance dependence within 3 months prior to screening evaluation (patient with a positive drug screen at screening may be included provided use does not lead to a diagnosis of substance dependence and patient consents to abstain from illegal drugs at any time during the study)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Measurement of implicit and explicit learning through cognitive testing over a period of 7 days | 7 days
  The cognitive data will be summarized and summary statistics calculated (including mean, standard deviation, median, minimum, and maximum values) for each experiment and participants group.

SECONDARY OUTCOMES:
Incidence of Adverse Events | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Duffel, Belgium